CLINICAL TRIAL: NCT03798548
Title: Brief Cognitive Behavioral Therapy for Patients Undergoing Transcatheter Aortic Valve Replacement: A Randomized Controlled Trial
Brief Title: Brief CBT for Patients Undergoing TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, William Fearon, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 32178
Record Dates: First submitted 2019-01-03; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Depression, Anxiety
Keywords: CBT; Brief Therapy; Bedside Intervention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Brief Bedside CBT versus Treatment As Usual
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Bedside CBT (Experimental)
  Interventions: Behavioral: Brief Bedside CBT
- Treatment As Usual (No Intervention)

INTERVENTIONS:
Behavioral: Brief Bedside CBT — 4 sessions of CBT including psychoeducation about TAVR and how mood can impact recovery in cardiac patients, discussion of patients' expectations and any concerns. Teaching and practice of cognitive restructuring and behavioral goal setting techniques for a healthy recovery.
  Arms: Brief Bedside CBT

SUMMARY:
Adult patients scheduled to undergo TAVR were randomized to receive brief bedside cognitive behavioral therapy for depression/anxiety or treatment as usual.

DETAILED DESCRIPTION:
Depression and anxiety are common symptoms in patients undergoing cardiac surgery and associated with increased cardiac morbidity and decreased functional status. Cognitive behavioral therapy (CBT) has been shown to be an effective intervention to treat these symptoms after cardiac surgery, but has not yet been studied in patients undergoing less invasive cardiac procedures such as Transcatheter Aortic Valve Replacement (TAVR). This study will examine the effect of CBT on symptoms of anxiety and depression in patients undergoing TAVR.

The CBT protocol was loosely structured on the Managing Depression and Anxiety using Education and Skills (MADES) protocol described in Dao and colleagues (2011). The current intervention was designed to address the needs of individuals who may develop anxiety or depression symptoms post-TAVR. The CBT intervention consisted of four 30 to 60-minute bedside treatment sessions with a trained clinician while the participant was hospitalized for TAVR.

Main outcome measures were self-reported symptoms of depression and anxiety as measured by the Beck Depression Inventory-II and State Trait Anxiety Inventory Form Y1. Secondary outcomes included health related quality of life and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age and older
2. Voluntary participation
3. Informed consent obtained
4. Patients with severe aortic stenosis and high surgical risk who are undergoing TAVR

Exclusion Criteria:

1. Current psychiatric instability (eg., suicidality, schizophrenia, bipolar disorder, active alcoholism or substance abuse)
2. Severe cognitive impairment, i.e. dementia
3. Life threatening co-morbidities
4. Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Score on Beck Depression Inventory II (BDI-II) | An average of 3 days post TAVR Procedure, 1-Month Follow Up
  21-item self-report questionnaire with good reliability and validity in assessing symptoms of depression. Total score range 0-63 with higher scores indicating a worse outcome. Total BDI-II scores are interpreted as follows, 0-13: minimal, 14-19: mild, 20-28: moderate, 29-63: severe. In this study, a score of 14 or greater, and 20 or greater, were used define subpopulations with significant symptoms of depression on the BDI-II.

SECONDARY OUTCOMES:
Change from Baseline Score on State Trait Anxiety Inventory Form YI (STAI-YI) | An average of 3 days post TAVR Procedure, 1-Month Follow Up
  20-item self-report questionnaire with good internal consistency and construct validity in assessing symptoms of anxiety. Total score range 20-80 with higher scores indicating a worse outcome. The recommended cutoff score for clinically significant anxiety is 39 but a recent validity study of anxiety disorders in cardiac patients found ≥ 40 as an optimal cutoff score for screening the presence of an anxiety disorder. In this study, a score of 40 or greater, and 46 or greater, were used to define subpopulations with significant symptoms of anxiety on the STAI-Y1.
Change from Baseline Score on Minnesota Living With Heart Failure Questionnaire (MLHFQ) | 1-Month Follow Up
  21-item self-report questionnaire designed to measure the effects of heart failure and treatments for heart failure on and individual's quality of life. Total score range 0-105. The total score is considered a measurement of heart failure severity as indicated by its adverse effect on the respondent's life over the past month. In this study, the MLHFQ total score was used as a continuous measure of heart failure related quality of life. Higher scores indicate a worse outcome.
Change from Baseline Score on 12-Item Short Form Health Survey (SF12v2) | 1-Month Follow Up
  An abbreviated version of the 36-item Short Form Health Survey, which is a well-established measure assessing dimensions of mental and physical health. In this study, PCS and MCS summary scores were used as continuous measures of health-related quality of life. Scoring procedures involve computer-based scoring algorithms to calculate two summary scores, the physical component summary score (PCS) and mental component summary score (MCS), on a scale from 0 to 100 with a mean of 50 ± 10 that is normally distributed according to the adult U.S. population. Higher scores indicate a better outcome.

REFERENCES:
- [Background] Dao TK, Youssef NA, Armsworth M, Wear E, Papathopoulos KN, Gopaldas R. Randomized controlled trial of brief cognitive behavioral intervention for depression and anxiety symptoms preoperatively in patients undergoing coronary artery bypass graft surgery. J Thorac Cardiovasc Surg. 2011 Sep;142(3):e109-15. doi: 10.1016/j.jtcvs.2011.02.046. Epub 2011 May 28. PMID 21621227